CLINICAL TRIAL: NCT02620566
Title: Evaluation of Anesthesia Profile in Pediatric Patients After Inguinal Hernia Repair With Caudal Block or Local Wound Infiltration
Brief Title: Caudal Block vs Local Wound Infiltration for Hernia Repair in Children
Acronym: CBvsLWI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Clinic for Anesthesia Reanimation and Intensive Care Mother Theresa (Other)
Responsible Party: Principal Investigator, Aleksandra Gavrilovska-Brzanov MD Msc., Principal Investigator, University Clinic for Anesthesia Reanimation and Intensive Care Mother Theresa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCTOARICED1
Record Dates: First submitted 2015-09-20; First posted 2015-12-03 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Anesthesia
Keywords: caudal block; local wound infiltration; hernia repair

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacain -Caudal (Active Comparator): Single shot Caudal Block will receive Group C with 1ml per kg Bupivacain 0,25%.
  Interventions: Procedure: Bupivacain- Caudal
- Bupivacain- Local (Active Comparator): Single shot Local Infiltration will receive Group L with 0,2ml per kg Bupivacain 0,25%.
  Interventions: Procedure: Bupivacaine- Local

INTERVENTIONS:
Procedure: Bupivacain- Caudal — Bupivacain for caudal blocks, Group C received 1 ml kg of 0.25% (maximum volume 20 ml).
  Other Names: Caudal block
  Arms: Bupivacain -Caudal
Procedure: Bupivacaine- Local — Bupivacain for Local Wound Infiltration Group L received 0,2 ml kg 0,25% (maximum volume 4 ml).
  Other Names: Local Wound Infiltration
  Arms: Bupivacain- Local

SUMMARY:
To our knowledge there is still no study comparing the local wound infiltration by itself without ilio-inguinal and ilio-hypogastric nerve block and caudal anesthesia. The aim of this study was to evaluate anesthesia and recovery profile in pediatric patients after inguinal hernia repair with caudal block (CB) or local wound infiltration (LWI).

DETAILED DESCRIPTION:
Total of 80 children aged 6 month to 7 years of ASA physical status I or II, undergoing unilateral hernia repair will be enroled in the study. One group will receive caudal block (CB) and the other group will receive local wound infiltration (LWI).

Group CB will receive 1ml kg 0,25% bupivacaine and group LWI will receive 0,2 ml kg 0,25% bupivacaine. Data taken will than be analyzed and interpreted. Postoperative pain will be assess using the Children's Hospital of Eastern Ontario Pain Scale (CHEOPS, 0-10)(8) and the Faces Legs Activity Cry Consolability tool (FLACC, 0-10)(9) at 30 min and 1, 2, and 3 h after operation. The time to first supplemental oral acetaminophen demand (first acetaminophen time) was defined as the time from the end of surgery to the first registration of more than 4 on both CHEOPS and FLACC by the investigator. Twenty-four hours after surgery, reports of delayed side-effects and demands for rescue acetaminophen from the child will be gathered. The investigator, who will be blind to the treatment group, will document these data with the medical records.

ELIGIBILITY:
Inclusion Criteria:

* 6 month to 7 years
* ASA physical status I or II
* undergoing unilateral hernia repair

Exclusion Criteria:

* history of developmental delay or mental retardation
* type I diabetes
* known or suspected coagulopathy
* known allergy to any local anesthetic
* known congenital anomaly of the spine
* signs of spinal anomaly or infection at the sacral or inguinal region

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to First Analgesic Requirement | 24 hours
  The time to first supplemental oral acetaminophen demand (first acetaminophen time) was defined as the time from the end of surgery to the first registration of more than 4 on both CHEOPS and FLACC by the investigator. At t0. 30 min postoperative; t1 1h postoperative; t2 2h postoperative; t3 3h posoperative; t4 6h posoperative; t5 12h posoperative; t6 24h postoperative

SECONDARY OUTCOMES:
The total number of oral acetaminophen | The number of analgesic received for the period of 24 hours
  Total number of analgesic requirement

OTHER OUTCOMES:
Postoperative Pain | 30 minutes postoperative, 1 hour postoperative, 2 hour postoperative, 3 hour postoperative, 6 hour postoperative , 12 hours postoperative, 24 post operative
  Postoperative pain was assessed using the Children's Hospital of Eastern Ontario Pain Scale (CHEOPS, 0-10).
Motor block | 30 minutes postoperative, 1 hour postoperative, 2 hour postoperative, 3 hour postoperative, 6 hour postoperative , 12 hours postoperative, 24 post operative
  Motor function was assessed using the following scale: 0, no motor block; 1, able to move legs; 2, unable to move legs.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Gavrilovska-Brzanov, MD. Msc, Principal Investigator — Mother Theresa University Clinical Center Skopje Macedonia
Locations (1):
- Uctoariced, Skopje, North Macedonia